CLINICAL TRIAL: NCT06781632
Title: Phase I Study Evaluating Safety, Pharmacokinetics, and Efficacy of a Combination Containing Ropivacaine, Clonidine, and Betamethasone (Ropiclobet, Batch:PL23001) for Sciatic Nerve Block in the Popliteal Region in Healthy Volunteers
Brief Title: Phase I Study of Ropivacaine, Clonidine, and Betamethasone Combination for Sciatic Nerve Block in the Popliteal Region
Acronym: RopiCloBet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PHARMAFINA (Industry)
Collaborators: MonitorCRO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF_001
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Nerve Block
Keywords: Ropivacaine; Clonidine; Betamethasone; Nerve Block
MeSH Terms: interventions — Ropivacaine; Clonidine; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nerve Block Arm (Experimental): Volunteers will undergo sciatic nerve block in the popliteal region using the combination drug Ropiclobet (Ropivacaine-Clonidine-Betamethasone)
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — Ropivacaine HCl - Betamethasone Sodium Phosphate - Clonidine HCl 5.0/0.4*/0.015 mg/mL (The solution contains 0.53 mg of betamethasone sodium phosphate, equivalent to 0.4 mg of betamethasone)
  Other Names: clonidine; betamethasone

SUMMARY:
This is a national, single-center, dose-escalation Phase I study to investigate the safety, pharmacokinetics, and efficacy of a combination containing Ropivacaine, Clonidine, and Betamethasone (Ropiclobet) in healty volunteers.

After screening and eligibility confirmation, at least 28 participants will receive a sciatic nerve block in the popliteal region with Ropiclobet, followed by pharmacokinetic assessments through blood sampling and monitoring of motor and sensory nerve blocks in the tibial and common peroneal nerves. Safety evaluations, including physical exams, vital signs, ECGs, and sedation scores, will be conducted throughout the study. sensory blocks resolve.

Participants will remain under observation for 48 hours post-procedure and will be discharged once motor and sensory blocks resolve. Follow-up visits will be conducted on Days 10 and 15 on an outpatient basis, with an end-of-study visit planned for Day 30.

The dose-escalation protocol involves administering 5 mL, 10 mL, 15 mL, and 20 mL doses to sequential groups of participants, with safety assessments performed after each dose level before proceeding.

DETAILED DESCRIPTION:
This is a national, single-center, dose-escalation Phase I clinical study designed to evaluate the safety, pharmacokinetics, and efficacy of a novel combination drug containing Ropivacaine, Clonidine, and Betamethasone, referred to as Ropiclobet, in healthy adult volunteers. The primary objective is to assess the safety of Ropiclobet when administered as a sciatic nerve block in the popliteal region. Secondary objectives include monitoring the drug's efficacy in inducing motor and sensory nerve blockade and evaluating its pharmacokinetic profile through.

The study will begin with the enrollment of a minimum of 28 healthy volunteers who meet the predefined eligibility criteria. Once deemed eligible, participants will receive a sciatic nerve block in the popliteal region using the investigational combination drug Ropiclobet. To investigate the pharmacokinetics of Ropiclobet, blood samples will be collected from each volunteer at carefully scheduled time points post-administration. These samples will be analyzed to determine the plasma concentrations of the three active components: Ropivacaine, Clonidine, and Betamethasone. Concurrently, effects of the drug will be evaluated by monitoring motor and sensory nerve blockades, specifically targeting the two primary branches of the popliteal nerve: the tibial nerve and the common peroneal nerve. Sensory blockade assessments will include tests for pin-prick and temperature sensations, while motor block evaluation will involve standardized clinical examinations.

Throughout the study, comprehensive safety monitoring will be conducted. This includes regular physical examinations, continuous vital sign measurements, electrocardiograms (ECGs), and the assessment of sedation levels. Volunteers will remain under observation in the Phase I clinic for at least 48 hours post-procedure. Discharge from the clinic will only occur after confirmation that both motor and sensory blocks have fully resolved. If the blocks persist beyond the 48-hour observation window, participants will be discharged no later than six hours following the resolution of the blockades. In addition to in-clinic assessments, follow-up evaluations will be performed on Days 10 and 15 on an outpatient basis, with a comprehensive end-of-study visit scheduled for Day 30. These visits aim to identify any delayed adverse effects and to ensure the complete recovery of participants.

The study's dose-escalation protocol involves four predefined dose levels of Ropiclobet: 5 mL, 10 mL, 15 mL, and 20 mL. Initially, 4 volunteers will receive a 5 mL dose for the sciatic nerve block. After a 48-hour observation period, detailed safety assessments will determine whether it is safe to proceed to the next dose level. If the safety profile of the 5 mL dose is deemed acceptable, an additional 8 volunteers will receive a 10 mL dose. This stepwise approach will continue with escalating doses of 15 mL and 20 mL, with safety evaluations conducted at each level before advancing to the subsequent dose. The final dose of 20 mL will only be administered if safety parameters remain within acceptable limits throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers based on the results of medical evaluation, including medical history, physical examination, neurological examination, laboratory tests, and cardiac monitoring, performed by the investigator.
* Between 18 and 45 years, male and female
* Provide a signed and dated written informed consent
* A negative pregnancy test at the screening visit for female volunteers with childbearing potential
* Negative alcohol breath test.
* Negative urine drug screening for addictive substances (amphetamine, barbiturates, benzodiazepines, cannabinoids, cocaine, opioids).
* Capable of completing all tests and evaluations related to the study.
* In the investigator's opinion, the volunteer must have the potential to comply with the study requirements.

Exclusion Criteria:

* Volunteers with hypersensitivity to local anesthesia/regional anesthesia.
* Volunteers with a known hypersensitivity to amide-based local anesthetics.
* Volunteers with chronic pain.
* Volunteers with neuromuscular diseases or peripheral neuropathy.
* Volunteers with bleeding disorders/coagulopathies.
* Volunteers with a history of motor or sensory loss in the lower extremities.
* Volunteers with a history of arrhythmia or seizures.
* Volunteers with renal or hepatic insufficiency.
* Volunteers diagnosed with diabetes.
* Volunteers with hereditary neuropathy.
* Volunteers with a body mass index (BMI) > 35 kg/m².
* Pregnant, breastfeeding, or women with a positive pregnancy test.
* Volunteers with skin infections or wounds at the injection site.
* Volunteers with clinically significant abnormalities in the ECG, such as rhythm, conduction, or morphology issues, or any abnormalities on a 12-lead ECG that could interfere with the interpretation of QTc interval changes (including normal ST-T wave morphology or left ventricular hypertrophy), as determined by the investigator or medical monitor, or those on chronic use of antiarrhythmic medications.
* Volunteers with clinically significant abnormalities in vital signs during screening, which may include:

  1. systolic blood pressure < 90 or > 140 mmHg,
  2. diastolic blood pressure < 50 or > 95 mmHg,
  3. heart rate < 45 or > 100 beats/min, measured three times at 5-minute intervals in a seated position.
* Volunteers with any condition (medical, psychological, social, etc.) that may impair their ability to comply with the study, as assessed by the investigator.
* Volunteers currently participating in another clinical study.
* Volunteers with a positive urine drug screening and/or alcohol test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Number of treatment-related adverse events assessed by NCI-CTCAE | From nerve block procedure to the end of study visit at 30 days
  The incidence of treatment-related adverse events, measured according to NCI-CTCAE criteria.
Number of treatment-related adverse events assessed by laboratory parameters | Before nerve block procedure, 24 and 48 hours after procedure, and during follow-up visits on Day 10, Day 15, Day 30
  The incidence of treatment-related adverse events based on hematological, and biochemical parameters
Number of treatment-related adverse events assessed by ECG | From nerve block procedure to discharge at 48 hours, and during follow-up visits on Day 10, Day 15, Day 30
  The incidence of treatment-related adverse events based on electrocardiography
Number of treatment-related adverse events assessed by physical examination and vital signs | From nerve block procedure to discharge at 48 hours, and during follow-up visits on Day 10, Day 15, Day 30
  The incidence of treatment-related adverse events based on physical examination and vital signs

SECONDARY OUTCOMES:
Pharmacokinetics (concentration analysis) | before the sciatic nerve block (at 0.hour) and post-block at 15, 30, and 45 minutes, and at 1, 2, 3, 4, 6, 8, 12, 18, 24, and 48 hours.
  The concentration-time profiles in plasma for each of the three active ingredients (Cmax)
Pharmacokinetics (concentration analysis) | before the sciatic nerve block (at 0.hour) and post-block at 15, 30, and 45 minutes, and at 1, 2, 3, 4, 6, 8, 12, 18, 24, and 48 hours.
  The concentration-time profiles in plasma for each of the three active ingredients (Area under curve)
Pharmacokinetics (concentration analysis) | before the sciatic nerve block (at 0.hour) and post-block at 15, 30, and 45 minutes, and at 1, 2, 3, 4, 6, 8, 12, 18, 24, and 48 hours.
  The concentration-time profiles in plasma for each of the three active ingredients (tmax)
Efficacy of ropiclobet assessed by onset of motor block | From nerve block procedure to the onset of motor block, up to 48 hours
  The time to the onset of complete motor block (in minutes or hours)
Efficacy of ropiclobet assessed by duration of motor block | From nerve block procedure to the resolution of the motor block, up to 48 hours
  The time of resolution of the motor block (in minutes or hours)
Efficacy of ropiclobet assessed by onset of sensorial block | From nerve block procedure to the onset of sensorial block, up to 48 hours
  The time to the onset of complete sensorial block (in minutes or hours)
Efficacy of ropiclobet assessed by duration of sensorial block | From nerve block procedure to the resolution of the sensorial block, up to 48 hours
  The time of resolution of the sensorial block (in minutes or hours)
Efficacy ropiclobet assessed by duration of motor and sensorial block | From onset of motor and sensorial block to the resolution, up to 48 hours
  Total motor and sensorial block time (in minutes or hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine Phase I and Clinical Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No